CLINICAL TRIAL: NCT00979407
Title: Immunological Equivalence Between GSK2340272A and GSK2340274A Influenza Vaccines in Adults Aged 18 to 60 Years
Brief Title: Study to Evaluate Immunological Equivalence Between Two Investigational Influenza Vaccines in Adults (H1N1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 113535
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2017-05

CONDITIONS: Influenza
Keywords: influenza infection; GSK Biologicals' influenza vaccine GSK2340272A and GSK2340274A
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- GSK2340272A GROUP (Experimental): Healthy male or female adults, between and including 18 to 60 years of age, who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
  Interventions: Biological: Influenza vaccine GSK2340272A
- GSK2340274A GROUP (Experimental): Healthy male or female adults, between and including 18 to 60 years of age, who received two doses of GSK2340274A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
  Interventions: Biological: Influenza vaccine GSK2340274A

INTERVENTIONS:
Biological: Influenza vaccine GSK2340272A — Two intramuscular injections at Day 0 and Day 21
  Arms: GSK2340272A GROUP
Biological: Influenza vaccine GSK2340274A — Two intramuscular injections at Day 0 and Day 21
  Arms: GSK2340274A GROUP

SUMMARY:
The primary purpose of the study is to assess the equivalence of the immune response elicited by two GSK Biologicals' adjuvanted influenza investigational vaccines (GSK2340272A and GSK2340274A) in adults aged 18 to 60 years. The second purpose of the study is to evaluate the safety and reactogenicity of these two vaccines.

DETAILED DESCRIPTION:
This Protocol Posting has been updated following Protocol Amendment 4, July 2010, leading to removal of one of the secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 60 years inclusive, at the time of the first vaccination.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Satisfactory baseline medical assessment by history and physical examination.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or multiple-user device
* Females of non-childbearing potential may be enrolled in the study.
* Female of childbearing potential may be enrolled in the study, if she:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of vaccination, and
* has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of an axillary temperature >= 37.5°C (99.5°F), or acute symptoms greater than "mild" severity on the scheduled date of first vaccination. NOTE: The subject may be vaccinated at a later date, provided symptoms have resolved, vaccination occurs within the window specified by the protocol, and all other eligibility criteria continue to be satisfied.
* Clinically or virologically confirmed influenza infection within 6 months preceding the study start.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Clinically or virologically confirmed influenza infection within 6 months preceding the study start.
* Chronic administration of immunosuppressants or other immune modifying drugs within 6 months of study enrolment or planned administration during the study period.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrolment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome.
* Administration of any vaccines within 30 days before vaccination.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* Pregnant or lactating female
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any conditions which, in the opinion of the investigator, prevents the subjects from participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 336 (Actual)
Dates: Start 2009-10-12 (Actual); Primary Completion 2009-11-09 (Actual); Study Completion 2010-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- France (3):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Poitiers
- Germany (3):
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Schmiedeberg, Saxony

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Launay O, Duval X, Fitoussi S, Jilg W, Kerdpanich A, Montellano M, Schwarz TF, Watanveerade V, Wenzel JJ, Zalcman G, Bambure V, Li P, Caplanusi A, Madan A, Gillard P, Vaughn DW. Extended antigen sparing potential of AS03-adjuvanted pandemic H1N1 vaccines in children, and immunological equivalence of two formulations of AS03-adjuvanted H1N1 vaccines: results from two randomised trials. BMC Infect Dis. 2013 Sep 16;13:435. doi: 10.1186/1471-2334-13-435. PMID 24041010
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 113535 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113535 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113535 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113535 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113535 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113535 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 336 subjects enrolled in the study, 2 subjects did not receive any vaccination.
Period: Overall Study
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Started | 167 | 167
Completed | 161 | 160
Not Completed | 6 | 7
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP | Total
Number analyzed (Participants) | 167 | 167 | 334
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.1 (11.65) | 39.7 (11.98) | 39.90 (11.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 77 | 164
  Male | 80 | 90 | 170
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African heritage / african american | 2 | 3 | 5
  Geographic ancestry: White - arabic / north african heritage | 0 | 3 | 3
  Geographic ancestry: White - caucasian / european heritage | 165 | 161 | 326

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The flu strain assessed was Flu A/CAL/7/09. The reference seropositivity cut-off value was greater than or equal to (≥) 1:10.
Time Frame: At Day 21
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity at Day 21, which included all evaluable subjects who received 1 vaccine dose and for whom assay results were available for antibodies against H1N1 antigen for the blood sample taken 21 days after the first vaccine dose.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 155 | 155
Titers | 383.6 [327.2 to 449.7] | 339.1 [285.4 to 403.0]

2. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies
Description: Seroconversion was defined as: For initially seronegative subjects [antibody titer below (<) 1:10 prior to vaccination], antibody titer greater than or equal to (≥) 1:40 after vaccination; For initially seropositive subjects (antibody titer ≥ 1:10 prior to vaccination), antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was A/California/7/2009 (H1N1)v-like influenza (Flu A/CAL/7/09).
Time Frame: At Days 21 and 42
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all evaluable subjects for whom 2 doses were taken and assay results were available for antibodies against H1N1 antigen for the blood sample taken 21 days after the first and second vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 155 | 155
Participants
  Flu A/CAL/7/09, Day 21 | 151 | 145
  Flu A/CAL/7/09, Day 42 | 154 | 153

3. Secondary Outcome: Number of SCR Subjects for HI Antibodies
Description: Seroconversion was defined as: For initially seronegative subjects [antibody titer below (<) 1:10 post to vaccination], antibody titer greater than or equal to (≥) 1:40 after vaccination; For initially seropositive subjects (antibody titer ≥ 1:10 prior to vaccination), antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was A/California/7/2009 (H1N1)v-like influenza (Flu A/CAL/7/09).
Time Frame: At Days 182 and 364
Population: The ATP cohort for persistence at Day 182 and 364 included all evaluable subjects who had received at least 1 dose of study/control vaccine, according to their treatment assignment during the primary vaccination course, and for whom assay results were available for antibodies against the study vaccine antigen component at Days 182 and 364.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 156 | 154
Participants
  Flu A/CAL/7/09, Day 182 | 144 | 141
  Flu A/CAL/7/09, Day 364: number analyzed (Participants) | 144 | 146
  Flu A/CAL/7/09, Day 364 | 109 | 106

4. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The flu strain assessed was Flu A/CAL/7/09. The reference seropositivity cut-off value was ≥ 1:10.
Time Frame: At Days 0 and 42
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all evaluable subjects for whom 2 doses were taken and assay results were available for antibodies against H1N1 antigen for the blood sample taken 21 days after the second vaccine dose.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 155 | 155
Titers
  Flu A/CAL/7/09, Day 0 | 9.5 [8.1 to 11.2] | 10.7 [9.1 to 12.7]
  Flu A/CAL/7/09, Day 42 | 599.8 [532.3 to 675.9] | 678.3 [599.3 to 767.6]

5. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 4
Time Frame: At Days 182 and 364
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 156 | 154
Titers
  Flu A/CAL/7/09, Day 182 | 202.5 [173.1 to 236.9] | 233.0 [196.0 to 276.9]
  Flu A/CAL/7/09, Day 364: number analyzed (Participants) | 144 | 146
  Flu A/CAL/7/09, Day 364 | 96.7 [81.2 to 115.2] | 107.6 [89.2 to 129.7]

6. Secondary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40, that usually is accepted as indicating protection.
Time Frame: At Days 0, 21 and 42
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all evaluable subjects who received 2 vaccine doses and for whom assay results were available for antibodies against H1N1 antigen for the blood sample taken 21 days after the first and second vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 155 | 155
Participants
  Flu A/CAL/7/09, Day 0 | 19 | 22
  Flu A/CAL/7/09, Day 21 | 155 | 151
  Flu A/CAL/7/09, Day 42 | 155 | 155

7. Secondary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: as for outcome 6
Time Frame: At Days 182 and 364
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 156 | 154
Participants
  Flu A/CAL/7/09, Day 182 | 151 | 150
  Flu A/CAL/7/09, Day 364: number analyzed (Participants) | 144 | 146
  Flu A/CAL/7/09, Day 364 | 121 | 121

8. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: GMFR was defined as the fold increase in serum HI geometric mean titers (GMTs) post-vaccination compared to pre-vaccination. The flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Days 21 and 42
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 155 | 155
Fold increase
  Flu A/CAL/7/09, Day 21 | 40.3 [33.2 to 49.0] | 31.6 [26.0 to 38.4]
  Flu A/CAL/7/09, Day 42 | 63.0 [52.2 to 76.1] | 63.2 [52.6 to 75.9]

9. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 8
Time Frame: At Days 182 and 364
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 156 | 154
Fold increase
  Flu A/CAL/7/09, Day 182 | 22.0 [18.5 to 26.1] | 21.7 [18.1 to 25.9]
  Flu A/CAL/7/09, Day 364: number analyzed (Participants) | 144 | 146
  Flu A/CAL/7/09, Day 364 | 11.0 [9.2 to 13.2] | 11.0 [9.1 to 13.3]

10. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects, who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 167 | 167
Participants
  Any Pain, Dose 1 | 148 | 144
  Grade 3 Pain, Dose 1 | 6 | 4
  Any Redness, Dose 1 | 25 | 19
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 32 | 29
  Grade 3 Swelling, Dose 1 | 2 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 162 | 162
  Any Pain, Dose 2 | 139 | 137
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 162 | 162
  Grade 3 Pain, Dose 2 | 5 | 4
  Any Redness, Dose 2: number analyzed (Participants) | 162 | 162
  Any Redness, Dose 2 | 18 | 17
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 162 | 162
  Grade 3 Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 162 | 162
  Any Swelling, Dose 2 | 17 | 21
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 162 | 162
  Grade 3 Swelling, Dose 2 | 1 | 0
  Any Pain, Across doses | 153 | 151
  Grade 3 Pain, Across doses | 8 | 6
  Any Redness, Across doses | 35 | 28
  Grade 3 Redness, Across doses | 0 | 0
  Any Swelling, Across doses | 36 | 36
  Grade 3 Swelling, Across doses | 2 | 0

11. Secondary Outcome: Number of Days With Solicited Local Symptoms
Description: The number of days with any solicited local symptoms reported during the solicited post-vaccination period.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Median (Inter-Quartile Range); unit: Days
Units Other Than Participants: Doses with the symptom
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 167 | 167
Number analyzed (Doses with the symptom) | 287 | 281
Days
  Pain, Post-Dose 1: number analyzed (Doses with the symptom) | 148 | 144
  Pain, Post-Dose 1 | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0]
  Pain, Post-Dose 2: number analyzed (Participants) | 162 | 162
  Pain, Post-Dose 2: number analyzed (Doses with the symptom) | 139 | 137
  Pain, Post-Dose 2 | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0]
  Pain, Overall/dose | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0]
  Redness, Post-Dose 1: number analyzed (Doses with the symptom) | 25 | 19
  Redness, Post-Dose 1 | 3.0 [2.0 to 6.0] | 3.0 [2.0 to 4.0]
  Redness, Post-Dose 2: number analyzed (Participants) | 162 | 162
  Redness, Post-Dose 2: number analyzed (Doses with the symptom) | 18 | 17
  Redness, Post-Dose 2 | 3.0 [2.0 to 4.0] | 2.0 [2.0 to 3.0]
  Redness, Overall/dose: number analyzed (Doses with the symptom) | 43 | 36
  Redness, Overall/dose | 3.0 [2.0 to 5.0] | 3.0 [2.0 to 4.0]
  Swelling, Post-Dose 1: number analyzed (Doses with the symptom) | 32 | 29
  Swelling, Post-Dose 1 | 3.0 [2.0 to 5.5] | 2.0 [1.0 to 5.0]
  Swelling, Post-Dose 2: number analyzed (Participants) | 162 | 162
  Swelling, Post-Dose 2: number analyzed (Doses with the symptom) | 17 | 21
  Swelling, Post-Dose 2 | 3.0 [2.0 to 4.0] | 2.0 [1.0 to 4.0]
  Swelling, Overall/dose: number analyzed (Doses with the symptom) | 49 | 50
  Swelling, Overall/dose | 3.0 [2.0 to 5.0] | 2.0 [1.0 to 4.0]

12. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, headache, joint pain at other location, muscle aches, shivering, sweating and fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination. Grade 3 symptom = general symptom that prevented normal everyday activities as assessed by inability to attend/do work or school, or required intervention of a physician/healthcare provider. Grade 3 fever = temperature > 39.0 °C and ≤ 40°C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 167 | 167
Participants
  Any Fatigue, Dose 1 | 60 | 55
  Grade 3 Fatigue, Dose 1 | 3 | 2
  Related Fatigue, Dose 1 | 54 | 54
  Any Headache, Dose 1 | 55 | 48
  Grade 3 Headache, Dose 1 | 4 | 2
  Related Headache, Dose 1 | 46 | 44
  Any Joint pain, Dose 1 | 37 | 38
  Grade 3 Joint pain, Dose 1 | 1 | 2
  Related Joint pain, Dose 1 | 33 | 37
  Any Muscle aches, Dose 1 | 57 | 81
  Grade 3 Muscle aches, Dose 1 | 3 | 4
  Related Muscle aches, Dose 1 | 55 | 79
  Any Shivering, Dose 1 | 34 | 24
  Grade 3 Shivering, Dose 1 | 0 | 2
  Related Shivering, Dose 1 | 32 | 24
  Any Sweating, Dose 1 | 13 | 14
  Grade 3 Sweating, Dose 1 | 1 | 1
  Related Sweating, Dose 1 | 12 | 14
  Any Temperature, Dose 1 | 2 | 5
  Grade 3 Temperature, Dose 1 | 1 | 2
  Related Temperature, Dose 1 | 2 | 5
  Any Fatigue, Dose 2: number analyzed (Participants) | 162 | 162
  Any Fatigue, Dose 2 | 61 | 60
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 162 | 162
  Grade 3 Fatigue, Dose 2 | 3 | 4
  Related Fatigue, Dose 2: number analyzed (Participants) | 162 | 162
  Related Fatigue, Dose 2 | 59 | 59
  Any Headache, Dose 2: number analyzed (Participants) | 162 | 162
  Any Headache, Dose 2 | 57 | 51
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 162 | 162
  Grade 3 Headache, Dose 2 | 2 | 3
  Related Headache, Dose 2: number analyzed (Participants) | 162 | 162
  Related Headache, Dose 2 | 53 | 46
  Any Joint pain, Dose 2: number analyzed (Participants) | 162 | 162
  Any Joint pain, Dose 2 | 34 | 47
  Grade 3 Joint pain, Dose 2: number analyzed (Participants) | 162 | 162
  Grade 3 Joint pain, Dose 2 | 5 | 4
  Related Joint pain, Dose 2: number analyzed (Participants) | 162 | 162
  Related Joint pain, Dose 2 | 33 | 45
  Any Muscle aches, Dose 2: number analyzed (Participants) | 162 | 162
  Any Muscle aches, Dose 2 | 64 | 71
  Grade 3 Muscle aches, Dose 2: number analyzed (Participants) | 162 | 162
  Grade 3 Muscle aches, Dose 2 | 4 | 2
  Related Muscle aches, Dose 2: number analyzed (Participants) | 162 | 162
  Related Muscle aches, Dose 2 | 63 | 70
  Any Shivering, Dose 2: number analyzed (Participants) | 162 | 162
  Any Shivering, Dose 2 | 37 | 35
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 162 | 162
  Grade 3 Shivering, Dose 2 | 5 | 4
  Related Shivering, Dose 2: number analyzed (Participants) | 162 | 162
  Related Shivering, Dose 2 | 37 | 32
  Any Sweating, Dose 2: number analyzed (Participants) | 162 | 162
  Any Sweating, Dose 2 | 24 | 16
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 162 | 162
  Grade 3 Sweating, Dose 2 | 4 | 2
  Related Sweating, Dose 2: number analyzed (Participants) | 162 | 162
  Related Sweating, Dose 2 | 23 | 15
  Any Temperature, Dose 2: number analyzed (Participants) | 162 | 162
  Any Temperature, Dose 2 | 11 | 8
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 162 | 162
  Grade 3 Temperature, Dose 2 | 2 | 3
  Related Temperature, Dose 2: number analyzed (Participants) | 162 | 162
  Related Temperature, Dose 2 | 11 | 8
  Any Fatigue, Across doses | 92 | 79
  Grade 3 Fatigue, Across doses | 6 | 5
  Related Fatigue, Across doses | 87 | 78
  Any Headache, Across doses | 83 | 73
  Grade 3 Headache, Across doses | 6 | 5
  Related Headache, Across doses | 74 | 69
  Any Joint pain, Across doses | 53 | 66
  Grade 3 Joint pain, Across doses | 5 | 5
  Related Joint pain, Across doses | 49 | 64
  Any Muscle aches, Across doses | 85 | 104
  Grade 3 Muscle aches, Across doses | 6 | 5
  Related Muscle aches, Across doses | 83 | 102
  Any Shivering, Across doses | 57 | 47
  Grade 3 Shivering, Across doses | 5 | 6
  Related Shivering, Across doses | 56 | 45
  Any Sweating, Across doses | 28 | 28
  Grade 3 Sweating, Across doses | 5 | 3
  Related Sweating, Across doses | 27 | 27
  Any Temperature, Across doses | 12 | 11
  Grade 3 Temperature, Across doses | 3 | 5
  Related Temperature, Across doses | 12 | 11

13. Secondary Outcome: Number of Days With Solicited General Symptoms
Description: The number of days with any solicited general symptoms reported during the solicited post-vaccination period.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Median (Inter-Quartile Range); unit: Days
Units Other Than Participants: Doses with the symptom
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 167 | 167
Number analyzed (Doses with the symptom) | 121 | 152
Days
  Fatigue, Post-Dose 1: number analyzed (Doses with the symptom) | 60 | 55
  Fatigue, Post-Dose 1 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 4.0]
  Fatigue, Post-Dose 2: number analyzed (Participants) | 162 | 162
  Fatigue, Post-Dose 2: number analyzed (Doses with the symptom) | 61 | 60
  Fatigue, Post-Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Fatigue, Overall/dose: number analyzed (Doses with the symptom) | 121 | 115
  Fatigue, Overall/dose | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Headache, Post-Dose 1: number analyzed (Doses with the symptom) | 55 | 48
  Headache, Post-Dose 1 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Headache, Post-Dose 2: number analyzed (Participants) | 162 | 162
  Headache, Post-Dose 2: number analyzed (Doses with the symptom) | 57 | 51
  Headache, Post-Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Headache, Overall/dose: number analyzed (Doses with the symptom) | 112 | 99
  Headache, Overall/dose | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Joint pain, Post-Dose 1: number analyzed (Doses with the symptom) | 37 | 38
  Joint pain, Post-Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Joint pain, Post-Dose 2: number analyzed (Participants) | 162 | 162
  Joint pain, Post-Dose 2: number analyzed (Doses with the symptom) | 34 | 47
  Joint pain, Post-Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Joint pain, Overall/dose: number analyzed (Doses with the symptom) | 71 | 85
  Joint pain, Overall/dose | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Muscle aches, Post-Dose 1: number analyzed (Doses with the symptom) | 57 | 81
  Muscle aches, Post-Dose 1 | 2.0 [2.0 to 3.0] | 2.0 [1.0 to 3.0]
  Muscle aches, Post-Dose 2: number analyzed (Participants) | 162 | 162
  Muscle aches, Post-Dose 2: number analyzed (Doses with the symptom) | 64 | 71
  Muscle aches, Post-Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Muscle aches, Overall/dose | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Sweating, Post-Dose 1: number analyzed (Doses with the symptom) | 13 | 14
  Sweating, Post-Dose 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Sweating, Post-Dose 2: number analyzed (Participants) | 162 | 162
  Sweating, Post-Dose 2: number analyzed (Doses with the symptom) | 24 | 16
  Sweating, Post-Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Sweating, Overall/dose: number analyzed (Doses with the symptom) | 37 | 30
  Sweating, Overall/dose | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Shivering, Post-Dose 1: number analyzed (Doses with the symptom) | 34 | 24
  Shivering, Post-Dose 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0]
  Shivering, Post-Dose 2: number analyzed (Participants) | 162 | 162
  Shivering, Post-Dose 2: number analyzed (Doses with the symptom) | 37 | 35
  Shivering, Post-Dose 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0]
  Shivering, Overall/dose: number analyzed (Doses with the symptom) | 71 | 59
  Shivering, Overall/dose | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0]
  Temperature, Post-Dose 1: number analyzed (Doses with the symptom) | 2 | 5
  Temperature, Post-Dose 1 | 3.0 [1.0 to 5.0] | 1.0 [1.0 to 1.0]
  Temperature, Post-Dose 2: number analyzed (Participants) | 162 | 162
  Temperature, Post-Dose 2: number analyzed (Doses with the symptom) | 11 | 8
  Temperature, Post-Dose 2 | 1.0 [1.0 to 1.0] | 2.0 [1.0 to 2.0]
  Temperature, Overall/dose: number analyzed (Doses with the symptom) | 13 | 13
  Temperature, Overall/dose | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0]

14. Secondary Outcome: Number of Subjects With Potential Immune-mediated Diseases (pIMDs)
Description: A pIMD was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration.
Time Frame: From Day 0 up to Day 42
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 167 | 167
Participants | 0 | 0

15. Secondary Outcome: Number of Subjects With pIMDs
Description: as for outcome 14
Time Frame: During the entire study period (from Day 0 up to Day 364)
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 167 | 167
Participants | 1 | 0

16. Secondary Outcome: Number of Subjects With Any Adverse Event of Special Interest (AESIs)
Description: An AESI was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration.
Time Frame: During the entire study period (from Day 0 up to Day 364)
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A GROUP | GSK2340272A GROUP
Number analyzed (Participants) | 167 | 167
Participants | 0 | 0

17. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 21 days after the first vaccination (Days 0 - 20) and 63 days after the second vaccination (up to Day 84)
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 167 | 167
Participants
  Any AE(s), Days 0-20 | 37 | 31
  Grade 3 AE(s), Days 0-20 | 3 | 1
  Related AE(s), Days 0-20 | 17 | 11
  Any AE(s), up to Day 84 | 68 | 71
  Grade 3 AE(s), up to Day 84 | 16 | 8
  Related AE(s), up to Day 84 | 20 | 20

18. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 up to Day 364)
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
Number analyzed (Participants) | 167 | 167
Participants | 9 | 11

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: within the 84-day (Days 0-83) post-vaccination period; SAEs: during the entire study period (from Day 0 up to Day 364).
Arm/Group | GSK2340272A GROUP | GSK2340274A GROUP
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/167
Serious Adverse Events (participants affected / at risk) | 9/167 | 11/167
Other Adverse Events (participants affected / at risk) | 157/167 | 159/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2340272A GROUP (N=167) | GSK2340274A GROUP (N=167)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Testicular injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2340272A GROUP (N=167) | GSK2340274A GROUP (N=167)
Arthralgia (Musculoskeletal and connective tissue disorders) | 53 (71) | 66 (85)
Chills (General disorders) | 57 (71) | 47 (59)
Erythema (Skin and subcutaneous tissue disorders) | 35 (43) | 28 (36)
Fatigue (General disorders) | 92 (121) | 79 (116)
Headache (Nervous system disorders) | 83 (120) | 80 (116)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 28 (37) | 28 (30)
Myalgia (Musculoskeletal and connective tissue disorders) | 85 (121) | 104 (152)
Nasopharyngitis (Infections and infestations) | 13 (15) | 9 (9)
Pain (General disorders) | 153 (287) | 151 (281)
Pyrexia (General disorders) | 12 (14) | 10 (11)
Rhinitis (Infections and infestations) | 9 (9) | 4 (4)
Swelling (General disorders) | 36 (49) | 36 (50)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.